CLINICAL TRIAL: NCT04994262
Title: The Effect on Thirst, Nausea-Vomiting, Hemodynamic Parameters, and Comfort Levels of Menthol Lozenge Applied After Extubation to Patients to Undergoing Cardiovascular Surgery
Brief Title: The Effect on Thirst, Nausea-Vomiting and Comfort Levels of Menthol Lozenge Applied After Extubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 21-14
Record Dates: First submitted 2021-05-05; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Nausea; Vomiting; Thirst
Keywords: Nausea; Vomiting; Menthol; Thirst; CABG
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients in the intervention group will be given a lozenge with menthol at the 30th, 60th and 90th minutes after extubation and it will be explained that they should be dissolved in the mouth without swallowing, and the patients will be kept under observation during this time.
  Thirty, 60, 90, and 120 minutes after extubation: Patients' thirst level and severity of nausea will be evaluated with the Visual Analogue Scale (VAS) and the presence of vomiting will be questioned. In addition, its physiological parameters will be recorded. These parameters will be evaluated just before the menthol lozenge application at the 30th, 60th and 90th minutes.
  Sixty, 120, 180, and 240 minutes after extubation: The amount and types of analgesic and antiemetic usage of the patients will be recorded.
  Second postoperative day: The comfort level of the patients will be evaluated using the General Comfort Scale Short Form.
  Interventions: Other: Menthol Lozenge
- Control Group (No Intervention): Patients in the control group will be followed up according to their routine clinical procedures. Since there is no procedure or intervention in the clinical procedures, only the patients will be followed up. Patients in the control group will be followed up with the same forms at the same time.
  Thirty, 60, 90, and 120 minutes after extubation: Patients' thirst level and severity of nausea will be evaluated with the Visual Analogue Scale (VAS) and the presence of vomiting will be questioned. In addition, its physiological parameters will be recorded.
  Sixty, 120, 180, and 240 minutes after extubation: The amount and types of analgesic and antiemetic usage of the patients will be recorded hourly.
  Second day after surgery: The comfort level of the patients will be evaluated and recorded using the General Comfort Inventory Short Form.

INTERVENTIONS:
Other: Menthol Lozenge — In the study, "Oka Menthol", a herbal lozenge produced by Otacı, will be used. Its formula contains: menthol 0.26%, eucalyptol 0.065%, thymol 0.0002%, camphor 0.0002%, anise oil, thyme oil, coltsfoot, marshmallow flower, bovine tail flower extracts, glucose and sucrose.
  Medical properties: Otacı Oka Menthol Pastil shows antibacterial and fungicidal properties with eucalyptol in its composition. Menthol is effective against local anesthetic, local antitussive and irritation. It also plays a mild analgesic role with camphor in its content. It has an antibacterial and antifungal effect with thymol, a phenolic antiseptic. Otaco Oka Menthol Pastilles also contain extracts of coltsfoot, cow's tail flower and marshmallow flower which are anti-irritant and expectorant.
  Arms: Intervention Group

SUMMARY:
It is reported that approximately 17.5 million people die worldwide each year due to cardiovascular diseases, including ischemic heart disease, cerebrovascular disease and rheumatic heart disease. The most preferred method in the treatment of coronary artery disease is Coronary Artery Bypass Graft (CABG) surgery. This procedure routinely requires general anesthesia and endotracheal intubation. Patients due to these practices often experience nausea-vomiting and thirst after extubation. It is stated that menthol application, which is a low cost, easy to apply and safe method, can be effective in the management of these complications. As a result of the literature review, there is no study evaluating the effectiveness of the menthol lozenge in quenching thirst after extubation and in the management of nausea and vomiting. In this study, it is aimed to develop methods that accelerate the postoperative recovery by proving the effect of oral menthol lozenge intake after extubation on thirst, nausea-vomiting, physiological parameters and comfort level in patients undergoing CABG surgery. The universe of this randomized controlled study was planned by Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital will create patients who underwent CABG surgery. His sample, on the same dates, was Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital will create a total of 118 patients hospitalized in the Cardiovascular Surgery (Postoperative) Intensive Care Unit and undergoing CABG surgery that meet the inclusion criteria. Participants will be divided into two equal groups as intervention (n = 59) and control (n = 59) groups. Patient Information Form, Intraoperative Patient Evaluation Form, Visual Analogue Scale (VAS) for evaluation of thirst and nausea-vomiting, Physiological Parameter Control Form, Analgesic-Antiemetic Use Control Form, General Comfort Scale Short Form will be used for data collection. The intervention group will be given a lozenge containing menthol orally at the 30th, 60th and 90th minutes after extubation. Thirst, nausea-vomiting, physiological parameters, analgesic and antiemetic consumption and comfort levels of all patients will be evaluated. The data obtained from the study will be analyzed with appropriate statistical methods using the SPSS for Windows 22.0 program (Statistical Package for the Social Sciences).

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of oral menthol lozenge administered after extubation on thirst, nausea-vomiting, physiological parameters and comfort level, as well as analgesic and antiemetic consumption in patients who underwent cardiovascular surgery. With this research, it is aimed to increase patient comfort by providing evidence of the effect of low-cost oral menthol lozenge intake on the feeling of thirst, nausea-vomiting, analgesic and antiemetic integration after extubation on physiological parameters.

Practices aimed at eliminating many problems such as thirst, sore throat, nausea and vomiting experienced in the early postoperative period positively affect the physical, psychospirical, environmental, sociocultural comfort of the patient and strengthen their health-oriented behaviors. It has been reported that there is a relationship between health-enhancing behaviors and providing comfort. It is observed that patients who undergo surgical procedures experience many problems in the postoperative period, their comfort level decreases and they are widely affected, from prolonged hospital stay to mortality. There are many studies in the literature aimed at accelerating the recovery in the perioperative process and increasing patient satisfaction.

Complications such as thirst and nausea and vomiting, which are seen in the postoperative period and can be quite disturbing by patients, can be overlooked in clinical observations. It is planned to prove the effectiveness of the use of low-cost and easy-to-apply menthol lozenge in the management of these complications. In the light of the literature review, menthol was found to be effective in gastrointestinal system disorders, pain management, and dehydration. The use of oral menthol containing lozenge in quenching thirst after extubation, in the management of postoperative nausea and vomiting, and in improving patient comfort, as well as analgesic-antiemetic consumption and evaluation of physiological parameters are the original value of this study.

The universe of the research was carried out by Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital will create patients who underwent CABG surgery. His sample, on the same dates, was Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital will create a total of 118 patients hospitalized in the Cardiovascular Surgery (Postoperative) Intensive Care Unit and undergoing CABG surgery that meet the inclusion criteria.

Sampling calculation was done with G Power 3.1.9.7 package program. Based on the VAS score averages in the study conducted by Aydın (2016), the sample that will represent the population was calculated as 0.05 significance level, the power of the study 80% and the effect size 0.46 (medium level) at the 95% confidence interval. As a result of the statistical analysis, it was calculated that the study should be carried out with a minimum of 118 patients, 59 in the experimental group and 59 in the control group.

t tests - Means: Difference between two independent means (two groups) Analysis: A priori: Compute required sample size Input: Tail(s) = One Effect size d = 0.4617784 α err prob = 0.05 Power (1-β err prob) = 0.80 Allocation ratio N2/N1 = 1 Output: Noncentrality parameter δ = 2.5080987 Critical t = 1.6580957 Df = 116 Sample size group 1 = 59 Sample size group 2 = 59 Total sample size = 118 Actual power = 0.8019408 Randomization Method: After obtaining the permission of the ethics committee, patients who meet the inclusion criteria in the study and who have received written informed consent to participate in the study will be divided into two groups in equal numbers with the computer-based randomization method.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65
* Undergoing elective coronary artery bypass graft surgery
* Extubated within the first 8 hours in the intensive care unit after CABG surgery
* Class ASA I, II and III
* Mallampati classification I and II
* Have no swallowing difficulties and Mann swallowing assessment score ≥95
* Glasgow Coma Scale with 15 points
* Patients who agree to participate in the study will be included.

Exclusion Criteria:

* Body Mass Index of 40
* Have a history of allergies
* Having severe nausea and vomiting at the time of application Illiterate
* Having communication problems
* Patients with psychiatric problems and using drugs will be excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) for Evaluating Thirst Level | Change from baseline (30 minutes) thirst level at 120 minutes after extubation.
  The VAS is 10 cm long and graded on a horizontal line.
  Thirst Score Comment:
  0-3 points Mild Thirst 4-6 points Moderate Thirst 7-10 points Severe Thirst
Visual Analogue Scale (VAS) for Evaluation of Nausea and Vomiting | Change from baseline (30 minutes) nausea and vomiting at 120 minutes after extubation.
  It is used to convert numerically non-measurable values into a numerical state. Interpretation of nausea severity score averages
  Nausea Severity Interpretation:
  0-1 No nausea 2-4 Mild nausea 5-7 Moderate nausea 8-10 Severe nausea
General Comfort Scale Short Form (GAS-SF) | This test will be applied on the second day after the surgery.
  The sc items), relaxation (9 items), and overcoming problems (10 items). In the evaluation of the scale consisting of positive and negative items, negative items are summarized with reverse coding. The lowest possible value of 1 indicates low comfort, and the highest value of 6 indicates high comfort.ale includes the sub-dimensions of relaxation, relaxation (9

CONTACTS AND LOCATIONS:
Locations (1):
- Selma CAN, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No